CLINICAL TRIAL: NCT06724588
Title: Systematic Analysis of Bacterial Multidrug Tolerance in Longitudinal Isolates of Patients That Are Prone to Developing Urinary Tract Infections
Brief Title: Analysis of Bacterial Multidrug Tolerance in Patients Prone to Urinary Tract Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: Natalie Verstraeten (Other)
Responsible Party: Sponsor-Investigator, Natalie Verstraeten, Dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S65007
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Patients with Recurrent or Chronic UTIs; Patients with a Suprapubic Catheter; Patients with a Nephrostomy Catheter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples, catheters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective observational study aimed at collecting bacterial isolates from patients with recurrent or chronic UTIs, or patients with suprapubic or nephrostomy catheters.

DETAILED DESCRIPTION:
In some cases, antibiotic therapy is not sufficient to clear bacterial infections. The reason for this is often a reduced sensitivity of the pathogens to the administered antibiotic. This sensitivity is largely determined by genetically encoded antibiotic resistance. In addition, bacterial populations also harbor a small fraction of phenotypic variants that are temporarily insensitive to the lethal effects of antibiotics. These so-called persister cells are formed by phenotypic transition from an antibiotic-sensitive 'normal' cell to an antibiotic-tolerant dormant state. On the other hand, persister cells can also return to the 'normal' state and resume growth, giving rise to the formation of a new population. Persistors represent an important but poorly understood clinical problem. For example, they play an underappreciated role in the failure of antimicrobial therapy in chronic infections. In addition, persisters contribute to the development of antibiotic resistance.

Little is known about how persistence evolves when bacteria are confronted with continuous or repeated antibiotic pressure. In silico predictions and previous in vitro work have shown that persister levels increase with frequent antibiotic exposure and that the period in the tolerant state is determined by the duration of treatment. We hypothesize that a similar evolutionary strategy occurs in vivo and that this contributes to the chronic nature of many infections. To support this hypothesis, we propose to collect longitudinal isolates from patients with recurrent or chronic UTIs. Since these patients visit the hospital at irregular and unpredictable time intervals, we will also collect isolates from patients with a suprapubic catheter. These patients do not necessarily suffer from chronic infections, but suprapubic catheters are usually colonized by microbial biofilms. We will also collect isolates from patients with a nephrostomy catheter. Similar to patients with suprapubic catheters, these patients visit the hospital regularly (± 6 weeks interval) for routine catheter changes and during these consultations, urine samples and catheter tips are easily collected. Furthermore, many of these patients are exposed to multiple antibiotic regimens (including, in the case of nephrostomy patients, high-dose cefazolin or ceftriaxone at the time of catheter change), creating a unique opportunity to study the evolution of antibiotic tolerance in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Who are older than 18y
* Who are of male or female sex
* Who suffer from recurrent or chronic infections with or without neurological disorders (spina bifida, MS, paraplegic patients)
* Who have or are planned to undergo the insertion of a suprapubic catheter
* Who have or are planned to undergo the insertion of a nephrostomy catheter

Exclusion Criteria:

* Who refused the planned treatment
* Who are known to have poor therapy compliance
* Who are pregnant
* Who did not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the ward or consultation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Collection of longitudinal bacterial strains to be used for fundamental research | Per patient, 20 samples will be collected at 6-week intervals.
  Urine samples and catheter tips will be collected following SOC procedures for diagnostic purposes, at each visit of the patient. Bacteria will be isolated and further studied.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided